CLINICAL TRIAL: NCT03471520
Title: Earplugs and Eye Masks Worn at Night to Reduce the Incidence of Delirium in General Medicine Inpatients
Brief Title: Earplugs and Eye Masks for Reducing Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00087770
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Delirium; Hospital Acquired Condition
MeSH Terms: conditions — Delirium; Iatrogenic Disease | interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Earplugs and eye masks (Experimental)
  Interventions: Behavioral: Earplugs and eye masks

INTERVENTIONS:
Behavioral: Earplugs and eye masks — Patients in this study will be given earplugs and eye masks to be worn during sleep

SUMMARY:
There has been some recent evidence to support the use of earplugs and eye masks to prevent delirium, but the existing studies have been small, have not been thoroughly replicated, and have only been conducted with intensive care unit (ICU) patients. Therefore, we propose to conduct a single-arm pilot study for an eventual single-blinded randomized controlled trial designed to assess the efficacy of earplugs and eye masks worn at night for prevention of delirium in a population of general medicine inpatients over the age of 65. The primary outcome will be incidence of delirium as measured by Confusion Assessment Method (CAM). In this pilot study, we will assess feasibility and will not perform any statistical comparisons. In the subsequent randomized controlled trial, we will be comparing the hazard rates on an intention-to-treat basis. Secondary outcomes will be exploratory and include length of stay, cost data, and use of pharmacologic interventions for sleep, delirium, or agitation. There are no physical risks and no cost to the subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to General Medicine (units 8100 and 8300 only) from the Duke University Hospital (DUH) Emergency Department
* Age >= 65

Exclusion Criteria:

* Admitted from outside hospitals, clinics (i.e., direct admissions), or transferred from another department
* Admitted as "observation" (i.e., expected length of stay < 2 nights)
* Admitted > 24 hours prior to time of enrollment
* Non-English-speaking patients will be excluded because a language barrier would introduce inaccuracy into the CAM measurement and for feasibility reasons (e.g., availability of translator services)
* Blind or deaf patients will be excluded because they are unlikely to benefit from the intervention, but sensory-impaired patients will be included
* Patients lacking decision-making capacity for whom no Legally Authorized Representative (LAR) is available
* Primary reason for admission "altered mental status", drug withdrawal, stroke, or seizure
* Patients for whom a withdrawal pathway has been preemptively initiated based on their substance use history (e.g., the alcohol withdrawal pathway order set or other as needed ("PRN") orders for the indication of withdrawal)
* Delirium present at time of enrollment
* Glasgow Coma Scale (GCS) < 10 at time of enrollment
* Enrolled in this trial during a previous admission (i.e., we will not resample)
* Enrolled in a separate trial this admission
* Contraindication to using earplugs or an eye mask (e.g., facial trauma or other safety concern)
* Significant fall risk per nursing assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | The first 5 days of patients' hospitalization
  Will be assessed using the CAM
Feasibility as measured by number of patients screened | 5 days
Feasibility as measured by number of patients ineligible | 5 days
Feasibility as measured by number of patients who decline to participate | 5 days
Feasibility as measured by number of patients who dropped out of the study | 5 days
Feasibility as measured by number of patients who wore the earplugs | 5 days
Feasibility as measured by number of patients who wore the eye masks | 5 days
Feasibility as measured by number of CAM assessment days | 5 days
Feasibility as measured by number of patients who successfully completed the study | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Juliessa Pavon, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States